### Official Title: Network-guided TMS in Early Alzheimer's Disease (NetTMS)

**NCT:** 04549155

IRB Document Date: 09/05/2024

Form M0345



Consent to Participate in a Research Study ADULT
Network TMS

### CONCISE SUMMARY

The purpose of this study is to explore network dynamics in the brain using MRI (magnetic resonance imaging) and TMS (transcranial magnetic stimulation), a non-invasive brain stimulation method, in older adults as a possible method to improve cognitive function. The study consists of 5 visits (ranging from 1 to 3 hours each). You will be compensated for your participation.

There are some risks involved in this study, such as a muscle-tension type headache and a rare risk of inducing a seizure. These and other risks will be discussed further in the consent form.

You are being asked to take part in this research study because you have either been referred to this study by your clinician, meet the inclusion criteria based on information from your medial record and visits to the Duke Neurology clinic, or are a member of another research study at Duke and have expressed interest in possibly participating in this study.

If you are interested in learning more about this study, please continue reading below.

Research studies are voluntary and include only people who choose to take part. Please read this consent form carefully and take your time making your decision. As your study doctor or study staff discusses this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. We encourage you to talk with your family and friends before you decide to take part in this research study. The nature of the study, risks, inconveniences, discomforts, and other important information about the study are listed below.

Please tell the study doctor or study staff if you are taking part in another research study.

A grant from the National Institutes of Health (NIH) will sponsor this study. Portions of Dr. Davis' salary and his research team's salaries will be paid by this grant.

### WHO WILL BE MY DOCTOR ON THIS STUDY?

If you decide to participate, Dr. Andy Liu will be your doctor for the study and will be in contact with your regular health care provider throughout the time that you are in the study and afterwards, if needed.

Simon W Davis, Ph.D. is conducting the study. A grant from the National Institutes of Health (NIH) will sponsor this study. Portions of Dr. Davis' salary and his research team's salaries will be paid by this grant.

DUHS |RB IRB NUMBER: Pro00106545 IRB REFERENCE DATE: 09/05/2024 IRB EXPIRATION DATE: 09/10/2025



### WHY IS THIS STUDY BEING DONE?

The purpose of this study is to explore how network dynamics in the brain interact to process information and how this processing can be changed and improved by an investigational non-invasive brain stimulation procedure called TMS. TMS has been approved by the Food and Drug Administration (FDA) as a treatment for depression, but in this study TMS is being used to investigate the impact it has on connectivity between certain regions of your brain, so therefore is considered "investigational." The word "investigational" means TMS is still being tested in research studies and is not approved by the FDA for these purposes. We are pairing TMS with fMRI (function magnetic resonance imaging) to maximize our understanding of how TMS impacts the brain's networks.

#### HOW MANY PEOPLE WILL TAKE PART IN THIS STUDY?

Approximately 55 people will take part in this study at Duke.

### WHAT IS INVOLVED IN THE STUDY?

If you agree to be in this study, you will be asked to sign and date this consent form. You will have the following tests and procedures to make sure that you are eligible:

- Psychiatric screening and medical history
- TMS and MRI safety screening
- Urine screening

The purpose of the urine test is to make sure you are not using any substance which could increase the risks of TMS. You may also be asked to provide a saliva sample obtained through cheek swab to test for risk factors for Alzheimer's Disease. This is a genetic test. Providing the saliva sample is optional and you may indicate your choice later in this consent form.

On Day 1, if you pass the screening procedure, you will be asked to fill out necessary forms and complete a series of tests for cognitive function.

On Day 2-5, you will have pictures of your brain taken using magnetic resonance imaging (MRI) while performing a computer task. MRI uses strong magnetic fields and radio waves to make pictures. Special pictures will be taken that provide information about the connectivity between the left and right halves of your brain. During this part of the study, you will lie on your back on a narrow bed that will be pushed into the MRI machine. The MRI technician will provide padding for your head and knees to make you more comfortable. If you are uncomfortable or feel pain because of lying down, tell the technician immediately. The technician will position your head inside a head tube, and the platform will be pushed into the MRI machine. You will hear a loud noise while the machine is collecting pictures. You will be able to communicate with the technician during the study using a microphone and speaker in the MRI machine. You may take a break at any time. You may stop your participation in this study at any time.



During the MRI scan you will complete a behavioral test, the Word Encoding task, in which you will see words of everyday objects and asked to respond using a keyboard. Then, in a later session, we will use your MRI data to identify a specific area to target with TMS. This session will last approximately 1 hour.

You will be introduced to transcranial magnetic stimulation (TMS) to allow you to find out what it is like. During this time, the study team will determine the proper strength of TMS to use in later visits. In this study, TMS will be used in a manner which is an investigational procedure, aimed at temporarily changing the way that a part of your brain works. The TMS equipment produces brief electrical currents that create a short-lived magnetic field. When the TMS equipment is held close to the head it can induce very small electric currents in the part of the brain that is closest to the coil. These currents are similar to the currents that the neurons in the brain produce when communicating with each other. By inducing these currents with the TMS, we can temporarily change the way that brain region functions, either making the region work harder or less hard.

Before applying TMS, the study team will determine what strength of stimulation to use for you by establishing your personal "motor threshold" – a measure of the excitability of the area of the human brain called the motor cortex. To establish this threshold, the study doctor or a member of the study staff will first place the stimulator over the part of your brain that controls the motor activity in your right hand. You will hear a clicking sound and feel a tapping sensation at your scalp. The stimulator will be adjusted to give just enough energy so that the motor region of the brain sends signals to your hand muscles, to make your hand twitch. The smallest amount of energy required to make your hand twitch is called your individual "motor threshold."

You will undergo a combined TMS-MRI session where you will complete the Encoding Task in the MRI scanner while receiving TMS. These sessions will take approximately 3 hours each.

#### HOW LONG WILL I BE IN THIS STUDY?

Your participation in this study will approximately 5 visits: including screening measures, MRI, and 3 sessions of TMS during MRI over the following weeks, allowing up to 1 year for participation.

You can choose to stop participating at any time without penalty or loss of any benefits to which you are entitled. However, if you decide to stop participating in the study, we encourage you to talk to your doctor first.

### WHAT ARE THE RISKS OF THE STUDY?

MRI Scanning:

There are no known long-term health risks from exposure to the magnetic fields and radio waves used to make MRI brain pictures. However, it is not assured that harmful effects will not be recognized in the future. Strong magnetic fields pose safety risks because they attract metals such as iron, and radio waves can interfere with medical devices such as pacemakers. It can be dangerous for people that have medical



devices, metal objects, or metal debris in their bodies to go into a MRI machine. This includes certain dyes found in some tattoos. It is also dangerous to bring loose metal objects into the room containing the MRI machine, because those objects may be pulled towards the magnet and could injure somebody in their way. For these reasons, you will be given an interview and questionnaire prior to this study to make sure that you can be safely scanned. You will be asked to leave all metal objects in lockers provided in the waiting room of the MRI center. You will also be asked to remove any jewelry and articles of clothing with metal inserts or clasps before entering the magnet room. In addition, the MRI scanner makes a loud buzzing noise that could affect your hearing. You will be provided with earplugs and/or headphones in order to protect your hearing. Please ask the study staff or MRI technician if you are unsure about these instructions.

The study involves entering a large room in which a magnet is present. You will be placed on a narrow bed and then slid into a small tunnel approximately 6 feet in length and 25 inches in diameter. You will be asked to lie still for about one hour on this bed. You will hear a loud machine-like noise. You may be asked to have a harmless monitoring device applied during the study. During the study, you can have voice contact and physical contact with someone in attendance if you desire. Some people feel anxious when confined by the small space of the MRI machine. If you feel anxious or uncomfortable inside the MRI machine, you can tell the study staff over the intercom and you will be removed immediately from the MRI machine.

### Incidental MRI Findings:

Medical specialists will not examine the research brain pictures. If you believe that you require a diagnostic MRI test, you should discuss your concerns with your doctor. The brain pictures obtained during this study are for research only and are not designed to search for any existing brain abnormalities. The study staff at Duke is not responsible for a failure to find any existing brain abnormalities. However, in the unlikely event that the technician or study staff collecting the scans notices something that appears abnormal, the technician will ask your permission to obtain an additional set of brain pictures that will be shown to a medically trained expert for clinical evaluation. The results of this evaluation will be provided to you at no charge. The decision to proceed with further examination or treatment based upon this evaluation lies solely with you. You will be responsible for any treatment that you undertake based upon this evaluation.

#### TMS:

The most serious known risk of TMS is seizure. TMS procedures are associated with a very low risk of seizures. Out of over 10,000 people given various forms of TMS to date, 16 people (less than 0.2%) have been reported to have had a seizure. TMS can produce a seizure when a series of pulses is given at high power and when repeated series of pulses are given extremely close together. This study will use only levels of TMS that are within safety guidelines. Levels of TMS that fall within the safety guidelines have not been associated with seizure in appropriately screened individuals. No seizures have occurred in normal volunteers with the dosage of TMS used in this study. To minimize this risk, we will medically screen you for any of the known characteristics that could lead to seizure. For example,



persons with epilepsy cannot participate in this study. You will be visually monitored during the TMS for any signs of seizure or muscle twitching. In spite of these precautions, there is a chance that you will experience a seizure. Should this occur, emergency facilities are available. If you have a seizure, you may require hospital admission and follow-up neurological evaluation. Having had a seizure may make it difficult for you to obtain medical insurance, future employment, and to drive. It is not known whether having had one seizure will make a person more prone to have future seizures. Should you have a seizure caused by TMS in this protocol, we will provide you with a letter documenting that the seizure was experimentally induced.

The most commonly reported side effect of TMS is a "muscle-tension" type headache. We expect that about three out of ten people may experience a headache with the types of TMS used in this study. We will make every effort to reduce any discomfort. If a headache occurs, it usually starts during or immediately after the TMS and lasts from minutes to hours after TMS. The headache usually goes away with standard over-the-counter pain medications. Neck pain may also occur. You may also experience some discomfort on your head where the coil is held. This is due to contraction of scalp muscles. Numbness of the face lasting for a short time has also been reported in rare instances that may last for several weeks after receiving the procedure. Syncope (fainting) is considered a rare side effect of TMS and has been reported in individuals who faint during blood draws. If you should experience syncope, you will be withdrawn from the study and have your blood pressure monitored until it returns to a healthy level.

The clicking noises produced by the TMS procedure are loud enough to be damaging to your ears. You will therefore be required to wear earplugs, provided by the staff. Additional side effects considered to be rare in TMS are dizziness, memory impairment, trouble concentrating, and acute mood changes. If these occur, these effects do not last long and will resolve without need for treatment. There may be other risks that are currently unknown. The long-term effects of rTMS are not known.

### **Optional Genetic Testing:**

**Participation in genetic studies**: The genetic studies described are for research purposes only. Therefore, you will receive no results from this study. It is not the purpose of this study to look for or provide you with any medical information or diagnoses relating to your present condition or any other disease or illness. The research tests are not being used as diagnostic tests for any disease or illness. Your participation in this study is not a substitute for your regular medical care or check-ups.

Potential Risks and the Genetic Information Non-Discrimination Act (GINA): There is a potential risk of loss of confidentiality. Every effort will be made to protect your confidential information, but this cannot be guaranteed. The genetic information obtained as a result of your participation in this research will not be included in your medical record. Information from which you may be personally identified will be maintained in a confidential, secure location at DUHS, accessible only by authorized members of the study team, and will not be disclosed to third parties except as described in this consent form, with your permission, or as may be required by law.

Form M0345



## Consent to Participate in a Research Study ADULT Network TMS

The Genetic Information Nondiscrimination Act (GINA) is a Federal law that will protect you in the following ways:

- Health insurance companies and group plans may not request genetic information from this research;
- Health insurance companies and group plans may not use your genetic information when making decisions regarding your eligibility or premiums;
- Employers with 15 or more employees may not use your genetic information when deciding to hire, promote, or fire you or when setting the terms of your employment. GINA does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. GINA also does not protect you against discrimination based on an already-diagnosed genetic condition or disease.

| If you would like to provide a saliva sample for future research studies, initial here. Your |
|---|
| sample will not contain any information that can be used to identify you. You acknowledge that you will |
| not be notified of any incidental findings, as your information will be de-identified in an effort to protect |
| your confidentiality. |

If you would not like to provide a saliva sample for future research studies, initial here. You are still welcome to participant in the other elements of this study, as discussed in this form.

### ARE THERE BENEFITS TO TAKING PART IN THE STUDY?

This study is not a diagnostic medical test and will be of no direct benefit to you. We hope that the information we collect in this study will improve our knowledge about the function of the human brain.

### WILL MY INFORMATION BE KEPT CONFIDENTIAL?

Participation in research involves some loss of privacy. We will do our best to make sure that information about you is kept confidential, but we cannot guarantee total confidentiality. Your personal information may be viewed by individuals involved in this research and may be seen by people including those collaborating, funding, and regulating the study. We will share only the minimum necessary information in order to conduct the research. Your personal information may also be given out if required by law.

As part of the study, results of your study-related laboratory tests, and procedures may be reported to **NIH** and its affiliates. In addition, your records may be reviewed in order to meet federal or state regulations. Reviewers may include representatives from the Food and Drug Administration (**FDA**), **NIH**, the Duke University Health System Institutional Review Board, and others as appropriate. If any of these groups review your research record, they may also need to review your entire medical record.

Study records that identify you will be kept confidential as required by law. Federal Privacy Regulations provide safeguards for privacy, security, and authorized access. Except when required by law or for your care, you will not be identified by name, social security number, address, telephone number, or any

DUHS RB
IRB NUMBER: Pro00106545
IRB REFERENCE DATE: 09/05/2024
IRB EXPIRATION DATE: 09/10/2025



other direct personal identifier in study records disclosed outside of Duke University Health System (DUHS). For records disclosed outside of DUHS, you will be assigned a unique code number. The key to the code will be kept securely at DUHS.

All the data recorded as part of this study are used for the purposes of this research study only. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by the federal privacy regulations. This information may be further disclosed by the sponsor of this study, the NIH. If disclosed by the sponsor, the information is no longer covered by the federal privacy regulations.

The study results will not be sent to your physician to include in your medical record. However, in case you experience a seizure, the study staff will urge you to notify your primary care physician about the incidence.

The Department of Health and Human Services (HHS) has issued a Certificate of Confidentiality to further protect your privacy. With this Certificate, the investigators may not disclose research information that may identify you in any Federal, State, or local civil, criminal, administrative, legislative, or other proceedings, unless you have consented for this use. Research information protected by this Certificate cannot be disclosed to anyone else who is not connected with the research unless:

- 1) there is a law that requires disclosure (such as to report child abuse or communicable diseases but not for legal proceedings);
- 2) you have consented to the disclosure, including for your medical treatment; or
- 3) the research information is used for other scientific research, as allowed by federal regulations protecting research subjects.

Disclosure is required, however, for audit or program evaluation requested by the agency that is funding this project or for information that is required by the Food and Drug Administration (FDA).

You should understand that a Confidentiality Certificate does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it. This means that you and your family must also actively protect your own privacy.

Finally, you should understand that the investigator is not prevented from taking steps, including reporting to authorities, to prevent serious harm to yourself or others.



All of the procedures and testing are being done only because you are in this study. The study results will **not** be provided to you OR sent to your physician.

The study results will be retained in your research record forever. Any research information in your medical record will also be kept indefinitely.

This information may be further disclosed by the sponsor of this study. If disclosed by the sponsor, the information is no longer covered by federal privacy regulations. If this information is disclosed to outside reviewers for audit purposes, it may be further disclosed by them and may not be covered by federal privacy regulations.

While the information and data resulting from this study may be presented at scientific meetings or published in a scientific journal, your name or other personal information will not be revealed.

Some people or groups who receive your health information might not have to follow the same privacy rules. Once your information is shared outside of DUHS, we cannot guarantee that it will remain private. If you decide to share private information with anyone not involved in the study, the federal law designed to protect your health information privacy may no longer apply to the information you have shared. Other laws may or may not protect sharing of private health information.

### WHAT ARE THE COSTS TO YOU?

There will be no costs to you for the research procedures.

### WHAT ABOUT COMPENSATION?

You will be paid \$20 per hour for participating in this study. This is to compensate you for your expenses related to participation (parking, gas, and time). The total amount of time required for participating in this study will be about 15 hours. Payments will be issued either via direct deposit within the Duke Unique ID system or by check form mailed to your home. Payment will be processed and sent for your receipt within a few weeks of your completion of the study.

Travel Reimbursement: Participants traveling a distance over 100 miles per day to attend sessions will be compensated for any mileage commuted over those 100 miles. Compensation will be at the federally mandated travel reimbursement rate up to \$200.

### WHAT ABOUT RESEARCH RELATED INJURIES?

Immediate necessary medical care is available at Duke University Medical Center in the event that you are injured as a result of your participation in this research study. However, there is no commitment by Duke University, Duke University Health System, Inc., or your Duke physicians to provide monetary compensation or free medical care to you in the event of a study-related injury.



For questions about the study or research-related injury, contact Dr. Davis at 919-668-2299 or the study doctor, Dr. Liu at 919-668-2879 during regular business hours. You can contact Dr. Davis at 919-943-7491 or Dr. Liu at 785-218-7574 after hours and on weekends and holidays.

### WHAT ABOUT MY RIGHTS TO DECLINE PARTICIPATION OR WITHDRAW FROM THE STUDY?

You may choose not to be in the study, or, if you agree to be in the study, you may withdraw from the study at any time. If you withdraw from the study, no new data about you will be collected for study purposes other than data needed to keep track of your withdrawal.

Your decision not to participate or to withdraw from the study will not involve any penalty or loss of benefits to which you are entitled, and will not affect your access to health care at Duke. If you do decide to withdraw, we ask that you contact Dr. Davis in writing and let him know that you are withdrawing from the study. His mailing address is Department of Neurology, Duke University Medical Center, Durham, NC 27710.

We will tell you about new information that may affect your health, welfare, or willingness to stay in this study. Dr. Davis may decide to take you off this study if you are unable to make your scheduled session appointments. If this occurs, you will be notified.

A description of this clinical trial will be available on <a href="https://www.clinicaltrials.gov/">https://www.clinicaltrials.gov/</a> as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this Web site at any time.

Availability/withdrawal of genetic samples: You will not have access to the sample once it is obtained. Samples may be stored indefinitely. If you decide to withdraw your permission to use your samples in this research project, please contact the Principal Investigator, Dr. Simon Davis, in writing and let him know you are withdrawing your permission for your samples to be stored and used for this or future research. His mailing address is simon.davis@duke.edu. At that time, we will ask you to indicate in writing if you want your unused samples destroyed or if your samples (with all identifying information removed that would link the sample to you) could be used in research. Data collected using your sample before your withdrawal will continue to be used as part of the study.

### WHOM DO I CALL IF I HAVE QUESTIONS OR PROBLEMS?

For questions about the study or a research-related injury, or if you have problems, concerns, questions or suggestions about the research, contact Dr. Davis at 919-668-2299 during regular business hours and at 919-599-1927 after hours and on weekends and holidays.

Form M0345



### Consent to Participate in a Research Study ADULT Network TMS

For questions about your rights as a research participant, or to discuss problems, concerns or suggestions related to the research, or to obtain information or offer input about the research, contact the Duke University Health System Institutional Review Board (IRB) Office at (919) 668-5111.

### STATEMENT OF CONSENT

"The purpose of this study, procedures to be followed, risks and benefits have been explained to me. I have been allowed to ask questions, and my questions have been answered to my satisfaction. I have been told whom to contact if I have questions, to discuss problems, concerns, or suggestions related to the research, or to obtain information or offer input about the research. I have read this consent form and agree to be in this study, with the understanding that I may withdraw at any time. I have been told that I will be given a signed and dated copy of this consent form."

| Signature of Subject | Date | Time |
|---------------------------------------|------|------|
| Signature of Person Obtaining Consent | Date | Time |